CLINICAL TRIAL: NCT04447170
Title: Comparison Between Laparoscopic and Open Repair of Perforated Gastroduodenal Peptic Ulcer
Brief Title: Laparoscopic Versus Open Repair of Peptic Ulcer Perforation
Acronym: LOREPUP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gianluca Costa (Other)
Responsible Party: Sponsor-Investigator, Gianluca Costa, Professor, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: I-Go-GIPS_2020_1
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Surgery; Emergencies; Peptic Ulcer Perforation
Keywords: Peptic ulcer perforation; Laparoscopy
MeSH Terms: conditions — Emergencies; Peptic Ulcer Perforation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laparoscopic repair: Patients undergoing laparoscopic treatment
  Interventions: Procedure: Simple repair or Graham technique
- Open repair: Patients undergoing open treatment

INTERVENTIONS:
Procedure: Simple repair or Graham technique — Simple suture with or without omental protective patch
  Groups: Laparoscopic repair

SUMMARY:
Although laparoscopic repair (LR) of perforated peptic ulcers (PPUs) has long been accepted, clinical evidence comparing LR versus open repair (OR) remains lacking. The aim of this study is to evaluate the feasibility, safety and outcome of laparoscopic gastric repair and compare it with the outcome open repair by relying on a propensity score matching statistical technique

DETAILED DESCRIPTION:
Despite the evolution of medical management of Gastroduodenal Peptic Ulcer (GPU), complications like bleeding and perforation are still not uncommon in clinical practice. According to the literature in average, 2-14% of peptic ulcers result in perforation, most 215 commonly occurring in females over the age of 60 and chronic NSAID, alcohol or tobacco users.

Management of perforated peptic ulcer entails resuscitation, pharmacotherapy and surgery.

Traditionally, suture with or without omental patch has been considered the 'gold standard' and still is. It is associated with shorter length of stay, lower transfusion needs and has lower morbidity as compared to gastrectomy. In 1992, it has been proposed that laparoscopy should be routinely considered in the management of perforated duodenal ulcer. Nowadays due to the advances in laparoscopic technique, many publications suggest that laparoscopic repair of perforated peptic ulcers could be a superior choice to open repair. These is linked with the advantages of laparoscopic surgery over open surgery such as reduced postoperative pain, lower wound infection rate, decreased length of hospital stay, and earlier functional recovery

ELIGIBILITY:
Inclusion Criteria:

* Patients surgically treated for benign peptic ulcer perforation

Exclusion Criteria:

* Age < 18 years
* Pregnant and breastfeeding women
* Malignant ulcer perforation
* Gastric resection
* Diagnostic laparoscopy/laparotomy with no further surgical procedures performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicenter italian national case-control study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
30-day Mortality Rate | 18 months
30-day Morbidity Rate | 18 months
  Morbidity defined by mean of the most used classification scoring system

SECONDARY OUTCOMES:
Conversion rate | 18 months
  Defined when a procedure was attempted via the minimally invasive approach but required an open incision to be completed
Calculation of Boey index | 18 months
  Calculation and evaluation of its predictive value for morbidity and mortality
Calculation of Mannheim Peritonitis Index | 18 months
  Calculation and evaluation of its predictive value for morbidity and mortality
Calculation of Shock index | 18 months
  Calculation and evaluation of its predictive value for morbidity and mortality
Calculation of Age-related shock index | 18 months
  Calculation and evaluation of its predictive value for morbidity and mortality
Operative time | 18 months
  The duration time of surgical step from in
  The duration of the surgical procedure
Calculation of Charlson Age-Comorbidity Index (CACI) | 18 months
  Calculation and evaluation of its predictive value for morbidity and mortality

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Policlinico San Pietro, Ponte San Pietro, Bergamo
  - Arcispedale S. Anna di Cona - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini di Roma, Rome, Lazio
  - Ospedale Cristo Re, Rome, Lazio
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale Civile di Adria, Adria, Rovigo
  - Cagliari University Hospital Monserrato, Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria Ospedale Riuniti Ancona, Ancona, The Marches
  - Ospedale della Misericordia Grosseto, Grosseto, Tuscany
  - Azienda Ospedaliera Pisana Policlinico Universitario Cisanello, Pisa, Tuscany
  - Ospedale San Giovanni Battista, Foligno, Umbria
  - Azienda Ospedaliera Santa Maria, Terni, Umbria
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome

REFERENCES:
- [Background] Cirocchi R, Soreide K, Di Saverio S, Rossi E, Arezzo A, Zago M, Abraha I, Vettoretto N, Chiarugi M. Meta-analysis of perioperative outcomes of acute laparoscopic versus open repair of perforated gastroduodenal ulcers. J Trauma Acute Care Surg. 2018 Aug;85(2):417-425. doi: 10.1097/TA.0000000000001925. PMID 29659470
- [Result] Ge B, Wu M, Chen Q, Chen Q, Lin R, Liu L, Huang Q. A prospective randomized controlled trial of laparoscopic repair versus open repair for perforated peptic ulcers. Surgery. 2016 Feb;159(2):451-8. doi: 10.1016/j.surg.2015.07.021. Epub 2015 Aug 19. PMID 26297055
- [Result] Siow SL, Mahendran HA, Wong CM, Hardin M, Luk TL. Laparoscopic versus open repair of perforated peptic ulcer: Improving outcomes utilizing a standardized technique. Asian J Surg. 2018 Mar;41(2):136-142. doi: 10.1016/j.asjsur.2016.11.004. Epub 2016 Dec 7. PMID 27955872